CLINICAL TRIAL: NCT06786910
Title: Effect on Cytokines IL-1ß, TNF-α, IL-4 and Total Bacterial Load of an Oral Topical Composition Comprising Olive Oil, Trymethylglycine and Xylitol: a Randomized Controlled Double-blind Clinical Trial Part of the Stop Dysbiosis Project (SDP)
Brief Title: Effect on Cytokines IL-1ß, TNF-α, IL-4, and Total Bacterial Load of a Composition Comprising Olive Oil, Trimethylglycine and Xylitol Delivered as a Toothpaste
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mucosa Innovations, S.L. (Industry)
Collaborators: University of Barcelona (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 03-2022
Record Dates: First submitted 2025-01-10; First posted 2025-01-22 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Inflammation; Interleukin-1beta; TNF-α; Cytokine Levels; BMI; Chronic Inflammatory Diseases; Dysbiosis; Overweight (BMI > 25)
Keywords: Inflammation; Cytokines; IL-1ß; TNF-α; BMI; Overweight; Dysbiosis; Chronic inflammatory diseases; Pro-inflammatory cytokines; olive oil, trimethylglycine and xylitol
MeSH Terms: conditions — Inflammation; Dysbiosis; Overweight | interventions — Toothpastes; Olive Oil; Betaine; Xylitol

STUDY DESIGN:
Intervention Model Description: Two toothpastes will be included in the study; one with the novel composition including olive oil, trimethylglycine and xylitol, and one without olive oil, trimethylglycine and xylitol. Both toothpastes, intervention and control, will be identical in aspect and flavour.
  Subjects are randomnly assigned: Researchers and participants will be blinded.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Toothpaste with olive oil, trimethylglycine and xylitol.
  Interventions: Other: Toothpaste with olive oil, trimethylglycine and xylitol
- Control group (Placebo Comparator): Toothpaste with identical flavour and aspect that experimental toothpaste but without olive oil, without trimethylglycine and without xylitol.
  Interventions: Other: Toothpaste without olive oil, trimethylglycine nor xylitol

INTERVENTIONS:
Other: Toothpaste with olive oil, trimethylglycine and xylitol — Composition comprising olive oil, trimethylglycine and xylitol, formulated as a toothpaste to be delivered topically onto the oral cavity 3 times a day during 1 month.
  Arms: Intervention group
Other: Toothpaste without olive oil, trimethylglycine nor xylitol — Composition without olive oil, without trimethylglycine and without xylitol, formulated as a toothpaste to be delivered topically onto the oral cavity 3 times a day during 1 month.
  Arms: Control group

SUMMARY:
The goal of this clinical trial is to learn if a novel composition comprising olive oil, trimethylglycine and xylitol, affects salivary levels of IL-1ß, TNF-α and IL-4 in a group of periodontally healthy, normal and overweight/pre-obese patients. The main question it aims to answer is if 1 month use of a composition under patent protection (patent pending, publication no. EP 4110321 A1 and US 2023/041103 A1) is able to reduce pro-inflammatory cytokines. The inflammatory background common to chronic inflammatory conditions is receiving the focus of research as it is thought to be originated in the overexpression of pro-inflammatory cytokines mainly IL-1ß and TNF-α considered today the link between the high burden of comorbidities associated to inflammation.

Researchers will compare the novel composition to a placebo (placebo toothpaste with same colour and flavour) to see if pro-inflammatory cytokine levels are reduced.

In a randomised double-blind controlled trial participants will be alleatorized to one of two groups, intervention or control. The composition will be delivered via toothpaste onto the oral mucosa in the intervention group while the control group will use a placebo toothpaste with the same characteristics but lacking the composition. All participants will be instructed to brush their teeth 3 times a day for one month without having had a dental cleaning before the start of the study.

DETAILED DESCRIPTION:
Barrier integrity plays a pivotal role in the homeostasis of the innate immune system. These barriers, their cells and networks, when intact and inhabited with an eubiotic microbiome, regulate immunity and inflammation, keeping the body in a state of homeostasis and balance with the outcome of health.

External pressure on mucosa and skin barriers from foreign substances and environmental circumstances, provides a changing ground for pro-inflammatory cytokine expression leading to what is known today as metabolic infection and systemic inflammation. Maintained pressure can exceed immune system control mechanisms, resulting in an ungoverned release of a variety of pro-inflammatory cytokines such as IL-1ß and TNF-α, that will further contribute to barrier breakage and to a state of immune dysregulation and inflammation. On the contrary, IL-4 has been ascribed both anti-inflammatory and pro-inflammatory properties.

Periodontal inflammation, the second most frequent contributor to systemic inflammatory load behind obesity, is an important factor upregulating salivary pro-inflammatory cytokines, and offers a practical model to address the complex crosstalk between inflammation and chronic inflammatory diseases.

STUDY DESIGN The current study will be a randomized controlled trial in periodontally healthy patients scheduled for a routine visit at the University of Barcelona (UB), Dental Hospital Barcelona University (HOUB), Bellvitge Campus.

Randomization and masking Patients will be randomly assigned by means of a random assignment sequence generated using Microsoft Office Excel 2019 (Microsoft Corporation, Washington, USA, 2013). A 1:1 distribution will be used to assign participants to either the Intervention Group (IG) or the Control Group (CG).

Intervention group will use an experimental toothpaste containing a novel composition comprising olive oil, trimethylglycine and xylitol. Control group will use a placebo toothpaste. Excipients will be common to both groups. All products will be packaged in white tubes with a label that will identify the number of patient. The product information allocated to each patient will be placed in a sealed envelope, exhibiting exclusively patient allocation number to maintain the integrity of the blinding process. Both, participants and operators will be masked to assignment.

Interventions Participants will be recruited during a routine visit to the University of Barcelona Dental Hospital. All participants from both groups will be attended at the dental clinic at the beginning and at the end of the study. During first visit baseline data will be recovered. Final visit will take place after one month for final data collection.

I. First Visit (T0):

Patients will be informed on the study details. Sex and age data will be recovered from medical history. No periodontal treatment, hygiene or profilaxis will be performed to avoid altering subgingival ecosystem. The following data will be recovered:

* Oral mucosa examination
* Decayed, missing and filled teeth (DMFT) index
* O'Leary Plaque Index
* Basic Periodontal Examination: Probing depth and clinical attachment loss
* Sialometry: Unstimulated and stimulated salivary flow were measured
* Salivary pH Unstimulated saliva will be used to cytokine analysis. Samples will be taken with sterile paper points inserted into the gingival sulcus of at least three teeth, preferably from 16, 22, 41, 47 for microbial analysis.

Participant´s weight and height will be recorded and body mass index (BMI) calculated to allow participants classification according to their nutritional status.

At the end of the visit, patients will receive their randomized assigned toothpaste and will be instructed to brush their teeth three times a day and refrain from using any other oral hygiene products. The second and final visit wil be scheduled after 1 month.

II. Second Visit (T1):

The procedure from first visit will be repeated, collecting the same data. Additionally, a visual analogue scale (VAS) will be provided for each patient who will rate ease of use, flavour, satisfaction, acceptance, preference, and recommendation from 0 to 10. Along the duration of the study and during the second and last visit, patients will be asked for any adverse or unwanted side effect. At this time, oral prophylaxis and dental cleaning will be performed.

Methodology:

Cytokine analysis Samples from unstimulated saliva will be sent immediately to the microbiology laboratory of UB Bellvitge Hospital. Samples will be centrifuged (14000 rpm, 10 min, 4ºC), and supernatants stored at -80ºC until determination of TNF-α, IL-1β, and IL-4 concentrations by enzyme linked immunosorbent assay (ELISA). Commercial kits (BioLegend ELISA MaxDeluxe Kit Human TNF, IL-1β e IL-4 and Human TNF, IL-1β e IL-4 Enhanced Sensitivity Flex test BD Cytometric Bead Array) will be used.

Additional analysis Microbiological analysis to assess subgingival total bacterial load will be performed with impregnated paper points that will be placed in a 2 ml cryotube and sent immediately to the microbiology laboratory of UB Bellvitge Hospital, where they will be frozen at -80ºC for further processing by quantitative polymerase chain reaction (real-time qPCR) using TaqMan assay. Total bacteria load, expressed as logarithmic units (log) of colony forming units per mL (cfu/ml), will be determined by amplifying 16S rRNA gene using universal procariotic primers.

Statistical analysis Sample size has been calculated using an α=0.05, a ß=0.2, and a 2-tailed significance level of 95%. Based on data from a pilot study testing the same composition.

Data were analysed with the SPSS Statistics software version 26. Categorical variables were described in frequency and percentage. Numerical variables, according to their distribution, in mean and standard deviation or median and minimum and maximum were expressed. Categorical variables were compared using the chi-square test for sex and t-student test for age. Numerical variables under study (inflammatory markers and bacterial load), having a non-normal distribution, were compared using non-parametric tests. To determine the differences of values between both groups (intervention and control) at the two times evaluated (T0: baseline; T1: after 1 month treatment) the Mann-Whitney U test was used for independent samples. To determine intragroup differences before and after the intervention/control, Wilcoxon's signed range test was used for related samples. A p<0.05 value was considered statistically significant.

For analyzing if there were intragroup differences in salivary flow, Fisher's test for independent samples and the McNemar test for related samples were used. The analysis was limited to two categories of the variable: "Normal" or "Low" (including both "Low" and "Very Low"). Regarding effect size calculation for primary outcomes, since the variables did not follow a normal distribution, non-parametric tests were used. The effect size, represented as r-value was calculated using the absolute value of the Z statistic obtained from the Wilcoxon or Mann-Whitney test, divided by the square root of the sample size (i.e., the number of paired values for related samples or the sum of sample sizes for independent samples).

ELIGIBILITY:
Inclusion Criteria:

* patients attending to a routinary control visit at the University of Barcelona Dental Hospital (HOUB) over 18 years of age;
* who give their informed consent to participate in the study;
* do not have associated medical pathology in ASA III and IV.

Exclusion Criteria:

* patients who do not wish to participate in the study;
* allergic to the components of the toothpaste;
* on active antibiotic treatment or having received antibiotic treatment within the past seven days;
* patients presenting pain or acute infections will be excluded as well as ASA III and IV; -
* patients with diabetes and BMI>40 and severe periodontitis will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2022-06-13 (Actual); Primary Completion 2022-09-15 (Actual); Study Completion 2022-09-15 (Actual)

PRIMARY OUTCOMES:
Changes in salivary IL-1ß levels. | T0 refers to the time at which baseline measurements are taken. T1 refers to 30 days.
  Differences between IL-1ß levels before and after the use of the assigned toothpaste for intervention and for control group.
Changes in salivary TNF-α levels. | T0 refers to the time at which baseline measurements are taken. T1 refers to 30 days.
  Differences between TNF-α levels before and after the use of the assigned toothpaste for intervention and for control group.
Changes in salivary IL-4 levels. | T0 refers to the time at which baseline measurements are taken. T1 refers to 30 days.
  Differences between IL-4 levels before and after the use of the assigned toothpaste for intervention and for control group.
Comparison of changes in IL-1ß levels between intervention and control groups. | T0 refers to the time at which baseline measurements are taken. T1 refers to 30 days.
  Each group will show a IL-1ß level at baseline and a IL-1ß level after 1 month use of the assigned toothpaste. Sense and magnitude of the changes observed for the intervention group will be compared with the changes observed for the control group.
Comparison of changes in TNF-α levels between intervention and control groups. | T0 refers to the time at which baseline measurements are taken. T1 refers to 30 days.
  Each group will show a TNF-α level at baseline and a TNF-α level after the use of the assigned toothpaste. Sense and magnitude of the changes observed for the intervention group will be compared with the changes observed for the control group.
Comparison of changes in IL-4 levels between intervention and control groups. | T0 refers to the time at which baseline measurements are taken. T1 refers to 30 days.
  Each group will show a IL-4 level at baseline and a IL-4 level after the use of the assigned toothpaste. Sense and magnitude of the changes observed for the intervention group will be compared with the changes observed for the control group.

SECONDARY OUTCOMES:
Changes in subgingival total bacterial load. | T0 refers to the time at which baseline measurements are taken. T1 refers to 30 days.
  Differences between subgingival total bacterial load at baseline and after the use of the assigned toothpaste for each of both groups.
Clinically assessed parameters at baseline and after the use of the assigned toothpaste. | T0 refers to the time at which baseline measurements are taken. T1 refers to 30 days.
  Bleeding on probing and plaque index, both expressed as percentage, at baseline and after the use of the assigned toothpaste for both groups.
Comparison of changes in cytokine levels, due to the use of the assigned toothpaste, between intervention and control group in patients with BMI>25. | T0 refers to the time at which baseline measurements are taken. T1 refers to 30 days.
  Assessment of cytokine levels at baseline and after 1 month use of the assigned toothpaste will be performed. Sense and magnitude of the changes observed for the intervention group will be compared with the changes observed for the control group for each cytokine in patients with BMI>25.

OTHER OUTCOMES:
Patient reported outcome measures of flavour, satisfaction, acceptance, preference and recommendation to use with the use of a visual analogue scale. | T1 refers to 30 days.
  Patients assessment of ease of use, flavour, satisfaction, acceptance, preference and recommendation to use with a visual analogue scale ranging from 0 to 10, being 10 the best result.

CONTACTS AND LOCATIONS:
Overall Officials: José López-López, Principal Investigator — Barcelona University
Locations (1):
- University of Barcelona, L'Hospitalet de Llobregat, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Dinarello CA, van der Meer JW. Treating inflammation by blocking interleukin-1 in humans. Semin Immunol. 2013 Dec 15;25(6):469-84. doi: 10.1016/j.smim.2013.10.008. Epub 2013 Nov 23. PMID 24275598
- [Background] Hajishengallis G, Chavakis T. Inflammatory memory and comorbidities. Clin Transl Med. 2022 Jul;12(7):e984. doi: 10.1002/ctm2.984. No abstract available. PMID 35839318